CLINICAL TRIAL: NCT04277065
Title: Short Outcomes Between Bulldog vs. Cotton Tourniquet in Laparoscopic Hepatectomy
Brief Title: Bulldog vs. Cotton Tourniquet in Laparoscopic Hepatectomy for Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: hui hou (Other)
Responsible Party: Sponsor-Investigator, hui hou, Director of the hepatobiliary surgery department, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Laparoscopic Liver Resection; Vascular Occlusion; Tourniquet
Keywords: Laproscopic hepatectomy; Bulldog; Vascular occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulldog tourniquet in laparoscopic Hepatectomy (Experimental): The bulldog tourniquet , a reusable vessel occlusion instrument forblocking the liver inflow-blood in laparoscopic liver resection, was uniformly employed in all patients randomized to Bulldog laparoscopic hepatectom group in the present study.
  Interventions: Procedure: BULLDOG ,A Useful Vascular Occlusion Tourniquet In Laparoscopic Liver Resection
- cotton tourniquet in laparoscopic Hepatectomy (Active Comparator): The cotton tourniquet ,a reusable vessel occlusion instrument for blocking the liver inflow-blood in laparoscopic liver resection
  Interventions: Procedure: cotton tourniquet

INTERVENTIONS:
Procedure: BULLDOG ,A Useful Vascular Occlusion Tourniquet In Laparoscopic Liver Resection — Bulldog is an effectively performed approach for vascular occlusion during laparoscopic hepatectomy than traditional Pringle manuever.
  Arms: Bulldog tourniquet in laparoscopic Hepatectomy
Procedure: cotton tourniquet — cotton tourniquet
  Arms: cotton tourniquet in laparoscopic Hepatectomy

SUMMARY:
LLR was applied for tumors located at the lower edge and lateral segments of the liver that could be resected more easily than posterosuperior segments. With the development of technology and the growing experience of hepatobiliary surgeons, LLR has been expanded to major liver resections, anatomical resections, and donor hepatectomies by skilled surgeons. However, postoperative mortality, mobility and recovery of liver function are associated with major blood loss which is always the main cause of conversion to laparotomy and remains a challenge for surgeons. Pringle first described the method to arrest the hepatic hemorrhage by compression of the porta hepatis and this procedure was widely spread as well as in laparoscopic feild currently. Here, we described a new modified of Pringle maneuver using Bulldog to block vascular during LLR, and compared its effects with traditional pringle maneuver.

DETAILED DESCRIPTION:
With the innovations of laparoscopic technique and specialized equipment , laparoscopic liver resection became the dominating resection surgery approach. December of 2014, laparoscopic hepatectomy was carried out in our department, extracorporeal Pringle maneuver has been applied in most laparoscopic liver resections which need to block the hepatic inflow, cotton tape was the frequently used tourniquet. We used to blocked the hepatic inflow by extracorporeal Pringle maneuver method with cotton tape for its validity , softness and no visible damages for vessel, but it was always difficult for clamping in a two-dimensional view to encircle the hepatoduodenal ligament , and it delayed operation time for freshmen. Bulldog has been widely used in urinary surgery for vascular occlusion, but bulldog in hepatic surgery has rarely been mentioned, this is the first report to formally demonstrate the clinical application in hepatic surgery. However, it is not clear that whether the bulldog for vascular occlusion is useful and easy to implement in laparoscopic hepatectomy. In this study, we will compare the cotton and the bulldog for vascular occlusion during laparoscopic hepatectomy

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent hepatectomy for benign or malignant neoplasm of the liver, and is suitable for laparoscopic liver resection
* Child-Pugh A without portal hypertension
* No portosystemic shunt
* No previous abdominal operation history
* American society of anesthesiology class(ASA): I or II
* Age 18 to 80

Exclusion Criteria:

* Additional intervention to the liver (Radio Frequent Ablation, Percutaneous Ethanol. Injection Therapy or others)
* Emergence hepatectomy
* Previous hepatectomy
* Combined operation for extrahepatic disease
* Vulnerable population (mental retardation, pregnancy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | intraoperative
  the volume of blood loss

SECONDARY OUTCOMES:
Liver functional recovery | up to 7 days after liver resection
  AST(glutamic oxalacetic transaminase, u/l)
Postoperative complication(Rates in different grades) | up to 30 days after liver resection
  According to The Clavien-Dindo Classification,https://www.assessurgery.com/clavien-dindo-classification/
Mortality rates | up to 30 days after liver resection
  the rate of postoperative death
Hospital duration after operation (days) | up to 30 days after liver resection
  the length of hospital stay
Operation time(min) | intraoperative
  the during of operation
Blood transfusion (times and units) | intraoperative
  intraoperative blood transfusion
the clamping and declamping time(s) | intraoperative
  the clamping and declamping time of using bulldog or cotton
Duration of abdominal drain (days) | up to 14 days after liver resection
  Duration of abdominal drain
Duration to first flatus (days) | up to 14 days after liver resection
  Duration to first flatus
Comfort questionnaire measures (GCQ) measures by Kolcaba | up to 30 days after liver resection
  GCQ measures by Kolcaba, download from http://www.thecomfortline.com/resources/cq.html
Intensive care unit stay(days) | up to 7 days after liver resection
  Intensive care unit stay in days
Liver functional recovery | up to 7 days after liver resection
  ALT(glutamic-pyruvic transaminase enzyme，u/l)
Liver functional recovery | up to 7 days after liver resection
  TB(total bilirubin，μmol/L)
Liver functional recovery | up to 7 days after liver resection
  ALB(albumin，g/L)
Liver functional recovery | up to 7 days after liver resection
  TP(total protein，g/L)

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd affiliated hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Background] Maehara S, Adachi E, Shimada M, Taketomi A, Shirabe K, Tanaka S, Maeda T, Ikeda K, Higashi H, Maehara Y. Clinical usefulness of biliary scope for Pringle's maneuver in laparoscopic hepatectomy. J Am Coll Surg. 2007 Dec;205(6):816-8. doi: 10.1016/j.jamcollsurg.2007.06.297. Epub 2007 Sep 18. No abstract available. PMID 18035269
- [Background] Dua MM, Worhunsky DJ, Hwa K, Poultsides GA, Norton JA, Visser BC. Extracorporeal Pringle for laparoscopic liver resection. Surg Endosc. 2015 Jun;29(6):1348-55. doi: 10.1007/s00464-014-3801-6. Epub 2014 Aug 27. PMID 25159645
- [Background] Ciria R, Cherqui D, Geller DA, Briceno J, Wakabayashi G. Comparative Short-term Benefits of Laparoscopic Liver Resection: 9000 Cases and Climbing. Ann Surg. 2016 Apr;263(4):761-77. doi: 10.1097/SLA.0000000000001413. PMID 26700223
- [Background] Rotellar F, Pardo F, Bueno A, Marti-Cruchaga P, Zozaya G. Extracorporeal tourniquet method for intermittent hepatic pedicle clamping during laparoscopic liver surgery: an easy, cheap, and effective technique. Langenbecks Arch Surg. 2012 Mar;397(3):481-5. doi: 10.1007/s00423-011-0887-3. Epub 2011 Dec 20. PMID 22183106
- [Background] Le B, Matulewicz RS, Eaton S, Perry K, Nadler RB. Comparative analysis of vascular bulldog clamps used in robot-assisted partial nephrectomy. J Endourol. 2013 Nov;27(11):1349-53. doi: 10.1089/end.2013.0367. Epub 2013 Oct 18. PMID 23895579
- [Background] Kim WJ, Kim KH, Shin MH, Yoon YI, Lee SG. Totally laparoscopic anatomical liver resection for centrally located tumors: A single center experience. Medicine (Baltimore). 2017 Jan;96(4):e5560. doi: 10.1097/MD.0000000000005560. PMID 28121916
- [Result] Ikeda T, Toshima T, Harimoto N, Yamashita Y, Ikegami T, Yoshizumi T, Soejima Y, Shirabe K, Maehara Y. Laparoscopic liver resection in the semiprone position for tumors in the anterosuperior and posterior segments, using a novel dual-handling technique and bipolar irrigation system. Surg Endosc. 2014 Aug;28(8):2484-92. doi: 10.1007/s00464-014-3469-y. Epub 2014 Mar 13. PMID 24622763